CLINICAL TRIAL: NCT00467428
Title: Efficacy and Safety of NS2359 in Adults With Attention Deficit Hyperactivity Disorder. A Randomised, Double-Blind, Placebo-Controlled Study
Brief Title: Efficacy and Safety of NS2359 in Adults With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroSearch A/S (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NS2359-001
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — GSK372475

INTERVENTIONS:
Drug: NS2359
Drug: Placebo

SUMMARY:
The purpose of the study is to investigate if NS2359 is effective in the treatment of ADHD in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of Attention Deficit Hyperactivity Disorder (ADHD), by DSM-IV, as manifested in clinical evaluation and confirmed by structured interview using the K-SADS-E adult ADHD module
* Patients with a CGI Global Severity (GS) score ≥4 (moderate impairment)
* The Patient provided written informed consent.
* Non-lactating women of childbearing potential that used adequate contraception (i.e. the use of oral contraceptives and practising a double-barrier form of birth control) and had a negative pregnancy test at screening. Women of no childbearing potential who had been postmenopausal for less than 2 years must have a negative pregnancy test at screening.

Exclusion Criteria:

* Any clinically unstable medical condition
* Clinically significant abnormal baseline laboratory values
* Mental retardation
* Organic brain disorders
* Non-febrile seizure disorder
* Patients with a history of an eating disorder including anorexia or bulimia nervosa
* Psychotic disorder of any type
* Patients with a HAM-D (17 item) >15
* Patients currently (within the past 6 months) known to abuse or to be dependent on any drug, including alcohol or a positive urine drug screen for cocaine, heroin, or marijuana
* Treatment with stimulants was prohibited within 1 week prior to randomisation
* Treatment with antipsychotics/neuroleptics was prohibited for 8 weeks prior to randomisation
* Treatment with monoamine oxidase inhibitors was prohibited for 8 weeks prior to randomisation
* Treatment with tricyclic antidepressants, histamines and selective serotonin reuptake inhibitors was prohibited for 4 weeks (fluoxetine for 6 weeks) prior to randomisation
* Treatment with benzodiazepines, anticonvulsants (for behaviour) and lithium for 2 weeks prior to randomisation
* Patients with a history of bipolar disorder
* Patients using any concurrent medication for the treatment of ADHD
* Patients that had previously participated in a NS2359 study
* Patients treated with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication
* Patients with a history of positive human immunodeficiency virus (HIV) test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2003-08; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
To investigate the efficacy of NS2359 in adult patients diagnosed with ADHD (predominantly inattentive, predominantly hyperactive/impulsive or combined) according to DSM-IV criteria.

SECONDARY OUTCOMES:
To investigate the safety and tolerability of NS2359 in adult ADHD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Thimothy Wilens, MD, Principal Investigator — Adult and Pediatric Psychopharmacology, Masschusetts General Hospial, Boston, US
Locations (1):
- Adult and Pediatric Psychopharmacology, Massachusetts General Hospital, Boston, Massachusetts, United States